CLINICAL TRIAL: NCT02064959
Title: HypOthermia for Patients Requiring Evacuation of Subdural Hematoma: a Multicenter, Randomized Clinical Trial
Brief Title: To Study the Effect of Early Cooling in Acute Subdural Hematoma Patients
Acronym: HOPES
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: interim analysis revealed it was futile, we would not reach an answer at N=60.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: The Vivian L. Smith Center for Neurologic Research (Other); Zoll Medical Corporation (Industry)
Responsible Party: Principal Investigator, Dong Kim, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-12-0762
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Subdural Hematoma, Traumatic
Keywords: Subdural Hematoma; Traumatic Brain Injury; Hypothermia
MeSH Terms: conditions — Hematoma, Subdural; Brain Injuries, Traumatic; Hypothermia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Hypothermia (Experimental): Hypothermia to 33°C
  Interventions: Device: Temperature management Zoll Intravascular Temperature Management device
- Normothermia (Active Comparator): standard care - normothermia (37°C)
  Interventions: Device: Temperature management Zoll Intravascular Temperature Management device

INTERVENTIONS:
Device: Temperature management Zoll Intravascular Temperature Management device

SUMMARY:
This randomized, prospective trial will study the effect of very early cooling in patients undergoing surgical evacuation of acute subdural hematomas (35°C prior to opening the dura followed by maintenance at 33°C for a minimum of 48h). Intravascular cooling catheters (Thermogard XP Device, Zoll) will be utilized to induce hypothermia or to maintain normothermia.

The primary objective is to determine if rapid induction of hypothermia prior to emergent craniotomy for traumatic subdural hematoma (SDH) will improve outcome as measured by Glasgow Outcome Scale-Extended (GOSE) at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Non-penetrating traumatic brain injury
* Glasgow Coma Scale (GCS) motor score ≤5 (not following commands)
* Estimated or known age 22-65 years
* Acute subdural hematoma requiring emergent craniotomy within 6 hours of initial injury
* Estimated time of injury to time to reach temp of 35°C<6 hrs

Exclusion Criteria:

* Total GCS = 3 and bilateral fixed and dilated pupils
* Following commands after an initial period of coma (GSC motor score of 6)
* Known pre-existing neurological deficit (e.g., previous traumatic brain injury (TBI), stroke)
* Concomitant spinal cord injury
* Arrival temperature is <35°C
* Hemodynamic instability (i.e., mean arterial pressure (MAP)<60 millimetres of mercury (mmHg) for 30 minutes)
* Active cardiac dysrhythmia resulting in hemodynamic instability
* Pregnancy
* Duret hemorrhage
* Prisoner or Ward of the State
* Known history of clotting disorder (e.g., heparin induced thrombocytopenia, pulmonary embolism/deep venous thrombosis)
* Injury to other body organ where hypothermia would be precluded because of bleeding risk (e.g., grade 3 liver laceration; bowel laceration; flail lung or international normalized ratio (INR) >1.4)
* Inability to obtain informed consent or utilize exception to informed consent for emergency research.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-03-22 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2019-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dong H. Kim, MD, Study Chair — The University of Texas Health Science Center, Houston
Locations (14):
- United States (5):
  - The University off Miami and Ryder Trauma Center, Jackson Memorial Hospital, Miami, Florida
  - Emory University, Atlanta, Georgia
  - University of Cincinnati, Cincinnati, Ohio
  - The University of Pittsburgh Medical Center and UPMC Presbyterian, Pittsburgh, Pennsylvania
  - The University of Texas at Houston Medical School and Memorial Hermann Hospital, Houston, Texas
- Japan (9):
  - Kurume University Hospital, Fukuoka
  - Saiseikai Fukuoka General Hospital, Fukuoka
  - Kagawa University Hospital, Kagawa
  - Nagasaki University Hospital, Nagasaki
  - Osaka Mishima Emergency Critical Care Center, Osaka
  - National Disaster Medical Center, Tokyo
  - Nippon Medical School Hospital, Tokyo
  - Nippon Medical School Tamanagayama Hospital, Tokyo
  - Yamaguchi University Hospital, Yamaguchi

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available.

REFERENCES:
- [Derived] Hergenroeder GW, Yokobori S, Choi HA, Schmitt K, Detry MA, Schmitt LH, McGlothlin A, Puccio AM, Jagid J, Kuroda Y, Nakamura Y, Suehiro E, Ahmad F, Viele K, Wilde EA, McCauley SR, Kitagawa RS, Temkin NR, Timmons SD, Diringer MN, Dash PK, Bullock R, Okonkwo DO, Berry DA, Kim DH. Hypothermia for Patients Requiring Evacuation of Subdural Hematoma: A Multicenter Randomized Clinical Trial. Neurocrit Care. 2022 Apr;36(2):560-572. doi: 10.1007/s12028-021-01334-w. Epub 2021 Sep 13. PMID 34518968

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were randomized and enrolled prior to evacuation of Subdural hematoma
Groups:
- Normothermia: Control, temperature maintained at 37°C
- Hypothermia: treatment group, temperature at 35°C at dura opening then 33°C > 48 hours
Period: Overall Study
Arm/Group | Normothermia | Hypothermia
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Normothermia: Control, temperature maintained at 37 degrees C
- Hypothermia: treatment group, temperature at 35 degrees C at dura opening then 33 degrees C > 48 hours
- Total: Total of all reporting groups
Arm/Group | Normothermia | Hypothermia | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 14 | 30
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] — under 18 years, between 18 and 65 years and greater than 65 years
  years | 41.2 (12.7) | 46.6 (15.1) | 43.9 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Participants: Female | 2 | 5 | 7
  Participants: Male | 14 | 11 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 13 | 11 | 24
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Population: Two regions enrolled subjects in this study
  participants
    United States | 12 | 13 | 25
    Japan | 4 | 3 | 7
Subdural hematoma present [Count of Participants; unit: Participants] | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Favorable Glasgow Outcome Score-Extended (GOS-E) at 6 Months Post Injury
Description: Participants were monitored for 6 months after injury, and GOS-E was scored as favorable (moderate disability to good recovery) or unfavorable (severe disability, vegetative state, or death) at 6 months post-injury.
Time Frame: 6 months post injury
Measure: Count of Participants; unit: Participants
Groups:
- Normothermia: Control, temperature maintained at 37 degrees °C
- Hypothermia: treatment group, temperature at 35 degrees °C at dura opening then 33 degrees °C > 48 hours
Arm/Group | Normothermia | Hypothermia
Number analyzed (Participants) | 16 | 16
Participants | 4 | 6

2. Secondary Outcome: Safety as Assessed by Number of Adverse Events Reported Per Participant
Description: Adverse events were graded according to the USDHHS Common Terminology Criteria for Adverse Events V4.0. Serious adverse events and pre-defined adverse events of interest that historically were known to be of concern with hypothermia treatment were selected to be monitored and reported regardless of grade. These included cardiac arrhythmias, thromboembolic events, pneumonia, bleeding or hemorrhage, intraoperative hemorrhage, infection (culture positive, e.g., blood stream infection, urinary tract infection, ventriculitis), device-related infection, and death. The number of adverse events per participant were compared between groups.
Time Frame: 6 months post injury
Measure: Median (Inter-Quartile Range); unit: number of adverse events per participant
Arm/Group | Normothermia | Hypothermia
Number analyzed (Participants) | 16 | 16
number of adverse events per participant | 4.500 [0.250 to 9.000] | 4.000 [2.000 to 7.750]

3. Secondary Outcome: Intensive Care Unit (ICU) Length of Stay
Time Frame: from ICU admission to ICU discharge (median of about 11 to 13 days)
Population: Data was not collected for one participant in the normothermia arm.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Normothermia | Hypothermia
Number analyzed (Participants) | 15 | 16
days | 11.390 [7.948 to 32.429] | 12.946 [9.234 to 17.719]

4. Secondary Outcome: Hospital Length of Stay
Time Frame: from hospital admission to hospital discharge (median of about 18 to 21 days)
Population: Data was not collected for one participant in the normothermia arm.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Normothermia | Hypothermia
Number analyzed (Participants) | 15 | 16
days | 18.243 [8.165 to 45.840] | 20.674 [17.769 to 29.784]

5. Secondary Outcome: Incidence of Cortical Spreading Depolarization
Time Frame: 6 months
Population: Data was not collected for this outcome measure.
Arm/Group | Normothermia | Hypothermia
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months post injury
Description: Adverse events with a grade of 3 or higher or predefined adverse events of interest(cardiac arrhythmia, thromboembolic event, pneumonia, pulmonary edema,bleeding/hemorrhage,infection(culture positive), device -related infection, Death)
Arm/Group | Normothermia | Hypothermia
All-Cause Mortality (participants affected / at risk) | 5/16 | 3/16
Serious Adverse Events (participants affected / at risk) | 10/16 | 11/16
Other Adverse Events (participants affected / at risk) | 10/16 | 12/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normothermia (N=16) | Hypothermia (N=16)
Anemia (Blood and lymphatic system disorders) | 6 (10) | 4 (10)
Elevated white blood cell count (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 1 (2) | 1 (2)
Tachycardia,agitation (Cardiac disorders) | 1 (1) | 0 (0)
Infection (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mesenteric ischemia with lactic acid disorder (elevated) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis, acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (5) | 4 (5)
Hypernatremia (Metabolism and nutrition disorders) | 4 (5) | 1 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 3 (4) | 1 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (6) | 2 (6)
Death (Nervous system disorders) | 5 (8) | 3 (8)
Epidural hematoma (Nervous system disorders) | 2 (2) | 0 (0)
hospital readmission,facial droop (Nervous system disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 2 (2) | 0 (0)
Elevated intracranial pressure (Nervous system disorders) | 2 (2) | 0 (0)
Intracranial Hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Muscle weakness upper limb (Nervous system disorders) | 0 (0) | 1 (1)
Neurological worsening (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 5 (6) | 1 (6)
Swelling and Hemorrhage during surgery (Nervous system disorders) | 1 (1) | 0 (0)
Worsening contusion (Nervous system disorders) | 1 (1) | 0 (0)
Urinary Tract infection (Renal and urinary disorders) | 2 (3) | 1 (3)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hospital readmission/chest wall hematoma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (9) | 5 (9)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sepsis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vascular Access Complication (Surgical and medical procedures) | 0 (0) | 1 (1)
hypotension (Vascular disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 5 (9) | 4 (9)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normothermia (N=16) | Hypothermia (N=16)
Anemia (Blood and lymphatic system disorders) | 4 (8) | 4 (8)
CPK Increased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphocyte decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 1 (3) | 2 (3)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (2) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Blood Bilirubin increased (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver dysfunction (Hepatobiliary disorders) | 0 (0) | 1 (1)
lipase increased (Investigations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 1 (2) | 1 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (3) | 2 (3)
Hypernatremia (Metabolism and nutrition disorders) | 2 (4) | 2 (4)
Hypokalemia (Metabolism and nutrition disorders) | 1 (3) | 2 (3)
hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (6) | 4 (6)
Wound Infection (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cranioplasty (Nervous system disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
seizure (Nervous system disorders) | 2 (4) | 2 (4)
Brain abscess (Nervous system disorders) | 0 (0) | 1 (1)
Meningitis (Nervous system disorders) | 0 (0) | 1 (1)
Neurological worsening (Nervous system disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (9) | 6 (9)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
scalp wound/infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Wound drainage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Replacement of catheter (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Thrombus(superficial) (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/59/NCT02064959/Prot_SAP_001.pdf